CLINICAL TRIAL: NCT01162993
Title: Effect of Spinal Cord Stimulation in Painful Diabetic Polyneuropathy: a Multicenter Randomised Controlled Trial (PDP Study)
Brief Title: Effect of Spinal Cord Stimulation (SCS) in Painful Diabetic Polyneuropathy
Acronym: PDP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 09-2-120
Record Dates: First submitted 2010-07-07; First posted 2010-07-15 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2016-10

CONDITIONS: Diabetic Neuropathies; Pain; Electric Stimulation Therapy
Keywords: Electric stimulation therapy; Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies; Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Cord Stimulation (Experimental): Spinal cord stimulation
  Interventions: Procedure: Spinal Cord Stimulation
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Procedure: Spinal Cord Stimulation — The intervention is spinal cord stimulation and will be used for 2 weeks trial stimulation. After clinical successful pain relief (≥50% relief of pain intensity on a weighted numeric rating scale (NRS) or a score of ≥6 on a seven-point Likert scale (1=very much worse; 7=very much improved) of the PGIC scale for pain and sleep) a definite spinal cord system will be implanted.
  Other Names: Medtronic leads and neurostimulator (CE mark 0123)
  Arms: Spinal Cord Stimulation

SUMMARY:
Rationale: Diabetic neuropathy is one of the most common complications of Diabetes Mellitus (DM). Pain is a common symptom of diabetic neuropathy, affecting 11-34% of patients suffering form DM. The burden of disease of painful diabetic polyneuropathy (PDP) is high for both the patient and society, due to significant pain levels, frequent co-morbidity, polypharmacy and significant health resource use. Spinal cord stimulation (SCS) has been used for over 30 years to treat neuropathic pain. Several small clinical studies have shown a beneficial effect of SCS on pain in PDP.

Objective: The primary objective of this study is to investigate whether SCS leads to clinically relevant (≥50%) pain relief in patients with moderate-to-severe PDP in the lower limbs after 6 months of treatment.

Secondary objectives to investigate 1) the effect of SCS on health related quality of life in PDP; 2) the effect of SCS on the quality of sleep in PDP; 3) the effect of SCS on mood in PDP; 4) the effect of SCS on blood glucose control in PDP; 5) the effect of SCS on large and small nerve fibre functions in PDP; 6) identifying predictive factors for success of SCS treatment of PDP; after 6 months 7) the effect of SCS on small fibre loss and regeneration in PDP; and 8) costs, cost-utility and cost-effectiveness after 12 months of treatment.

Study design: the study is a multi centre randomized controlled trial. Study population: Patients suffering from moderate-to-severe PDP in the lower limbs due to diabetes mellitus type 1 or type 2 as diagnosed by clinical symptoms (glove and stocking distribution).

Intervention: patients assigned to group 1 will receive spinal cord stimulation (SCS) and/or best (drug) treatment as possible, patients assigned to group 2 will receive best (drug) treatment as possible.

Main study parameters/endpoints: The main study parameter will be the mean pain intensity and/or maximal pain intensity during daytime and/or during night time as measured on a weighted NRS and/or a PGIC for pain and sleep measured on a 7-point Likert scale, after 6 months of treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: SCS related risks include: lead migration (14%), lead breakage (7%), implanted pulse generator migration (1%), loss of therapeutic effect, lost or unpleasant paresthesias (12%), infection or wound breakdown (10%), Pain at IPG incision site (12%), IPG pocket fluid collection (5%). Treatment-as-usual related risks are related to the medication used and do not increase due to participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe PDP in the lower limbs

  * The pain intended to treat has been present for more than 12 months
  * Previous treatment has been unsuccessful (insufficient pain relief and/or unacceptable side-effects) with drugs from the following drug categories:
  * Amitriptylin or an other tricyclic antidepressant and/or
  * Pregabalin (Lyrica®) or Gabapentin (Neurontin®) and/or
  * Duloxetine (Cymbalta®) and/or
  * Tramadol or strong opioids Patients were treated with 3 drugs from the above mentioned drug categories and followed the treatment algorithm for painful diabetic polyneuropathy according to Jensen. Starting dosage was based on individual patient characteristics. Each drug was tried for at least 3 weeks and dose was raised once, if possible. By insufficient pain relief and/or unacceptable side-effects, the drug treatment was stopped. Patients reached a steady state in medication use and it is not allowed to increase dosage during the study.
* Mean pain intensity during daytime and/or night time should be 5 or higher measured on a numeric rating scale (NRS). Pain during daytime will be scored 3 times per day during for 4 days according to Jensen.
* Patient's age is between 18 and 75 years.

Exclusion Criteria:

* The patient has had neuromodulation therapy during the month before the intake
* Neuropathic pain is most prevalent in the upper limbs (NRS>3)
* Neuropathy or chronic pain of other origin than diabetes mellitus (NRS> 3)
* Addiction: drugs, alcohol (> 5E / day) and/or medication

  * Drugs: cocaine, heroine, marihuana.
  * Alcohol: wine, beer, liquor (max 5E / day)
  * Medication: benzodiazepines.
* Insufficient cooperation from the patient (little motivation, understanding or communication)
* Blood clotting disorder, when using 2 or more different kinds of anti coagulation
* Immune deficiency (HIV-positive, corticosteroids with a dose equivalent to > prednisolone 10 mg, immunodepressive, etc.)
* Peripheral vascular disease without palpable peripheral pulses at both feet (inclusion is possible if pulses are absent, but ankle brachial index is between 0.7 and 1.2 in both feet)
* Active foot ulceration
* Life expectancy < 1 year
* Pacemaker
* Local infection or other skin disorders at site of incision
* Psychiatric problems potentially interfering with cooperation in the study
* Pregnancy
* Severe cardiac or pulmonary failure (> NYHA classification II)
* Unstable blood glucose control (change in HbA1c>1,0% in three months prior to inclusion)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured on a weighted NRS according to Jensen and a PGIC for pain measured on a 7-point Likert scale. | 6 months

SECONDARY OUTCOMES:
Effect SCS on health related quality of life, quality of sleep, mood, blood glucose control, large/small nerve fibre functions, predictive factors success of SCS treatment, small fibre loss/regeneration, cost-utility and cost-effectiveness | 6 and 12 months and 5 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van Kleef, Prf. Dr., Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - UMC St. Radboud, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg

REFERENCES:
- [Result] Tesfaye S, Watt J, Benbow SJ, Pang KA, Miles J, MacFarlane IA. Electrical spinal-cord stimulation for painful diabetic peripheral neuropathy. Lancet. 1996 Dec 21-28;348(9043):1698-701. doi: 10.1016/S0140-6736(96)02467-1. PMID 8973433
- [Result] Kumar K, Toth C, Nath RK. Spinal cord stimulation for chronic pain in peripheral neuropathy. Surg Neurol. 1996 Oct;46(4):363-9. doi: 10.1016/s0090-3019(96)00191-7. PMID 8876718
- [Result] de Vos CC, Rajan V, Steenbergen W, van der Aa HE, Buschman HP. Effect and safety of spinal cord stimulation for treatment of chronic pain caused by diabetic neuropathy. J Diabetes Complications. 2009 Jan-Feb;23(1):40-5. doi: 10.1016/j.jdiacomp.2007.08.002. Epub 2008 Apr 16. PMID 18413161
- [Result] Daousi C, Benbow SJ, MacFarlane IA. Electrical spinal cord stimulation in the long-term treatment of chronic painful diabetic neuropathy. Diabet Med. 2005 Apr;22(4):393-8. doi: 10.1111/j.1464-5491.2004.01410.x. PMID 15787662
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473
- [Derived] van Beek M, Geurts JW, Slangen R, Schaper NC, Faber CG, Joosten EA, Dirksen CD, van Dongen RT, van Kuijk SMJ, van Kleef M. Severity of Neuropathy Is Associated With Long-term Spinal Cord Stimulation Outcome in Painful Diabetic Peripheral Neuropathy: Five-Year Follow-up of a Prospective Two-Center Clinical Trial. Diabetes Care. 2018 Jan;41(1):32-38. doi: 10.2337/dc17-0983. Epub 2017 Nov 6. PMID 29109298
- [Derived] Slangen R, Faber CG, Schaper NC, Joosten EA, van Dongen RT, Kessels AG, van Kleef M, Dirksen CD. A Trial-Based Economic Evaluation Comparing Spinal Cord Stimulation With Best Medical Treatment in Painful Diabetic Peripheral Neuropathy. J Pain. 2017 Apr;18(4):405-414. doi: 10.1016/j.jpain.2016.11.014. Epub 2016 Dec 11. PMID 27965045
- [Derived] van Beek M, Slangen R, Schaper NC, Faber CG, Joosten EA, Dirksen CD, van Dongen RT, Kessels AG, van Kleef M. Sustained Treatment Effect of Spinal Cord Stimulation in Painful Diabetic Peripheral Neuropathy: 24-Month Follow-up of a Prospective Two-Center Randomized Controlled Trial. Diabetes Care. 2015 Sep;38(9):e132-4. doi: 10.2337/dc15-0740. Epub 2015 Jun 26. No abstract available. PMID 26116722
- [Derived] Slangen R, Schaper NC, Faber CG, Joosten EA, Dirksen CD, van Dongen RT, Kessels AG, van Kleef M. Spinal cord stimulation and pain relief in painful diabetic peripheral neuropathy: a prospective two-center randomized controlled trial. Diabetes Care. 2014 Nov;37(11):3016-24. doi: 10.2337/dc14-0684. Epub 2014 Sep 11. PMID 25216508